CLINICAL TRIAL: NCT05024968
Title: A Phase 2 Clinical Trial Evaluating the Efficacy and Safety of Sintilimab for Advanced Rare Cancers (SiARa Cancer Study) - Cancer of Unknown Primary (SiARa-CUP)
Brief Title: Sintilimab in Cancer of Unknown Primary
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Innovent Biologics (Suzhou) Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0902; NCI-2021-08870 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2021-08-19; First posted 2021-08-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Cancer of Unknown Primary Site
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (sintilimab) (Experimental): The study drug is sintilimab. The first dose of study treatment should start on Day 1 of Cycle 1. For the rest of the treatment cycles, the study treatment can be administered 3 day before or 3 days after the scheduled day of administration. Treatment can be delayed for up to 1 week if the administration day is on a holiday or if the subject is otherwise unavailable.
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — Given by IV

SUMMARY:
This is a Phase 2 clinical trial evaluating the efficacy and safety of sintilimab in subjects with CUP.

Up to 45 subjects with CUP will be enrolled. Subjects will be treated with sintilimab at 200 mg via intravenous (IV) administration on Cycle 1 Day 1. The treatment will repeat every 3 weeks until progressive disease (PD), intolerable toxicity, initiation of new anti-tumor therapy, withdrawal of consent, lost to follow-up, death, completion of therapy, or any other investigator-determined reasons for treatment discontinuation (whichever occurs first). Treatment will continue for a maximum period of 24 months (starting from the first dose).

During the trial, tumor imaging evaluation will be initially performed once every 9 weeks (± 7 days) and will be based on Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. After the completion or discontinuation of the study treatment, safety follow-up and survival follow-up will be performed.

Considering the rareness of the disease, the patient accrual rate is expected to be approximately 2 patients per month. The total study duration is expected to be between 24-27 months with 6-month follow up.

DETAILED DESCRIPTION:
Primary Objectives:

* To evaluate the safety and efficacy of sintilimab in subjects with CUP

Secondary Objectives:

* To evaluate the overall objective response rate (ORR) (investigator assessed), disease control rate (DCR), duration of response (DOR), progression-free survival (PFS), overall survival (OS) and Quality of Life (QOL) on sintilimab in subjects with CUP

Exploratory Objectives:

* To evaluate the correlation between biomarkers in tumor tissue and efficacy, including but not restricted to PD-L1 expression level, transcriptome sequencing, single-cell sequencing, and multicolor immunohistochemistry (IHC) analyses;
* To evaluate the correlation between biomarkers in peripheral blood and drug efficacy, including but not restricted to soluble PD-L1, circulating tumor DNA (ctDNA), and cytokine analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Has histopathologically confirmed unresectable, locally advanced, recurrent or metastatic CUP. Patients must have undergone standard work-up to attempt to identify the primary tumor prior to enrollment.
2. Is refractory or intolerant to at least one line of systemic chemotherapy. Patient ineligible for cytotoxic chemotherapy due to contraindications will be eligible.
3. Has an ECOG PS of 0 - 2.
4. Must be unsuitable for definitive treatment, such as definitive chemoradiotherapy and/or surgery. For subjects who have received (neo)adjuvant or definitive chemotherapy/chemoradiotherapy, time from the completion of last treatment to disease recurrence must be > 3 months.
5. Is able to provide archival or fresh tissues for correlative analysis with obtainable results.
6. Has at least one measurable lesion as per RECIST v1.1.
7. Has adequate organ and bone marrow functions, as defined below:

   * Complete blood count: absolute neutrophil count (ANC) ≥ 1.0 × 109/L, platelet (PLT) count ≥ 75 × 109/L, hemoglobin (HGB) ≥ 9.0 g/dL. Note: Subjects cannot receive blood transfusion, erythropoietin (EPO), or Granulocyte-colony stimulating factor (GSF) within 7 days prior to the blood collection.
   * Hepatic function: total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN in subjects without hepatic metastasis; TBIL ≤ 1.5 × ULN, ALT and AST ≤ 5 × ULN in subjects with hepatic metastasis.

   Exception: Patients with known Gilbert disease: serum bilirubin level ≤ 3 × ULN.
   * Renal function: urine protein < 2+ from random sample or < 1 g from 24-hour urine collection, and creatinine clearance rate (CrCl) ≥ 30 mL/min by Cockcroft-Gault formula:
   * Female: CrCl=((140-age)×weight(kg)×0.85)/(72×serum creatinine(mg/dL))
   * Male: CrCl=((140-age)×weight(kg)×1.00)/(72×serum creatinine(mg/dL))
8. Adequate coagulation function, defined as international normalized ratio (INR) ≤ 1.5 or prothrombin time (PT) ≤ 1.5 × ULN; if the subject is receiving anticoagulant therapy, the results of coagulation tests need to be within the acceptable range for anticoagulants.
9. Is expected to survive ≥ 12 weeks.
10. Subject (female subjects of childbearing age or male subjects whose partners are of childbearing age) must take effective contraceptive measures during the entire course of the trial and until 180 days after the last dose (see Section 4.3).
11. Is able to sign the informed consent form (ICF) and is able to comply with the scheduled follow-up visits and related procedures required in the protocol.

Exclusion Criteria:

1. Has received treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody, or any other antibody or drug that specifically targets T-cell co-stimulation or immune checkpoint pathways.
2. Is enrolled in another interventional clinical study. Current enrollment in an observational study (non-interventional) or in the follow-up phase of an interventional study is allowed.
3. Has received palliative therapy for a local lesion within 2 weeks prior to the first dose.
4. Has received systemic treatment with Chinese traditional medicines with anti-cancer indications or immunomodulators (including thymosins, interferons, and interleukins) within 2 weeks prior to the first dose of study treatment.
5. Has received systemic immunosuppressants within 2 weeks. Allowed are local use of glucocorticoids administered by nasal, inhaled, or other routes, and systemic glucocorticoids at physiological doses (no more than 10 mg/day of prednisone or equivalents), or glucocorticoids to prevent allergies to contrast media.
6. Has received a live attenuated vaccine within 4 weeks prior to the first dose of study treatment or is scheduled to receive live attenuated vaccine during the study period.

   Note: Seasonal inactivated influenza virus vaccines within 4 weeks prior to the first dose of study treatment are permitted, but attenuated influenza vaccines are not.
7. Has undergone major surgery (craniotomy, thoracotomy, or laparotomy) within 4 weeks prior to the first dose of study treatment or is scheduled to receive major surgery during the course of the trial.
8. Has any toxicity (excluding alopecia, events that are not clinically significant, or asymptomatic laboratory abnormalities) due to prior anti-tumor therapy that has not yet resolved to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 grade 0 or 1 prior to the first dose of study treatment.
9. Has known symptomatic central nervous system (CNS) metastasis or carcinomatous meningitis. Subjects with brain metastases who have received prior treatment can be enrolled if the disease is stable (no imaging evidence of PD for at least 4 weeks prior to the first dose of study treatment), there is no evidence of new brain metastases or progression of the existing metastatic lesion(s) upon repeated imaging, and corticosteroids have not been required for at least 14 days prior to the first dose of study treatment. Patients with carcinomatous meningitis are ineligible, regardless of whether the disease is clinically stable or not.
10. Has bone metastases and is at risk for paraplegia.
11. Has known active autoimmune disease requiring treatment or a previous autoimmune disease history within 2 years (subjects with vitiligo, psoriasis, alopecia, or Graves' disease not requiring systemic treatment, hypothyroidism only requiring thyroid replacement, or type I diabetes only requiring insulin can be enrolled).
12. Has a known history of primary immunodeficiency diseases.
13. Has a known active pulmonary tuberculosis.
14. Has a known history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation.
15. Is human immunodeficiency virus (HIV)-infected (has positive anti-HIV antibody).
16. Has an active or poorly controlled serious infections.
17. Has symptomatic congestive heart failure (NYHA Class II-IV) or symptomatic or poorly controlled arrhythmia.
18. Has uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg) despite standard treatment.
19. Had any arterial thromboembolic event within 6 months prior to enrollment, including myocardial infarction, unstable angina, cerebrovascular accident, or transient cerebral ischemic attack.
20. Has significant malnutrition, such as those requiring continuous parenteral nutrition ≥7 days. Allowed are those who received intravenous treatment for malnutrition that ended more than 4 weeks before the first dose of study treatment.
21. Has a history of clinically significant deep venous thrombosis, pulmonary embolism, or other serious thromboembolic events within 3 months prior to enrollment (having an implantable port or catheter-related thrombosis or incidental pulmonary embolism detected on scan without symptoms or superficial venous thrombosis is not considered to be a "serious" thromboembolisms).
22. Has uncontrolled metabolic disorders, non-malignant organ or systemic diseases, or cancer-related secondary diseases that may lead to higher medical risks and/or survival evaluation uncertainties.
23. Has severe pulmonary dysfunction.
24. Has hepatic encephalopathy, hepatorenal syndrome, or cirrhosis with Child-Pugh Class B or C.
25. Has bowel obstruction or history of any of the following diseases: inflammatory bowel disease, extensive bowel resection (partial colectomy or extensive small intestine resection accompanied with chronic diarrhea), Crohn's disease, or ulcerative colitis.
26. Has known acute or chronic active hepatitis B (positive HBsAg and hepatitis B (HBV) DNA viral load ≥ 103 copies/mL or > 200 IU/mL), or acute or chronic active hepatitis C (positive hepatitis C [HCV] antibody and detectable HCV RNA).
27. Has history of gastrointestinal (GI) perforation and/or fistula within 6 months prior to study enrollment (having a gastrostomy or enterostomy is allowed).
28. Has interstitial lung disease requiring corticosteroids.
29. Has history of other primary malignant tumors, excluding:

    * Malignant tumors that achieved a complete response (CR) at least 2 years prior to enrollment and expected to require no treatment during the trial.
    * Adequately treated nonmelanoma skin cancer or lentigo maligna with no sign of disease recurrence.
    * Adequately treated carcinoma in situ with no sign of disease recurrence.
    * Prostate cancer, CLL or other cancers where the indolent nature of tumor allows for and patient is under active surveillance.
30. Is pregnant or breastfeeding.
31. Has an acute or chronic diseases, psychiatric disorders, or laboratory abnormality that may lead to the following consequences: increased investigational drug-related risks, or interference with interpretation of trial results, or is otherwise considered ineligible for participating in the trial by the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-08-26 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Objective response rate (ORR) [Efficacy] | Within 4 cycles of treatment (1 cycles equals 28 days)

SECONDARY OUTCOMES:
Number of participants with Treatment-Emergent Adverse Events [Safety] | From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 1 year
Disease control rate (DCR) | Up to 2 years
Duration of response (DOR) | Time from response till progression, relapse/refractory, or death, assessed up to 2 years
Progression-free survival (PFS) | Time interval between treatment start until disease progression, relapse/refractory, or death due to any cause, assessed up to 2 years
Overall survival (OS) | Time interval between treatment start until death due to any cause, assessed up to 2 years
Quality of Life (QOL) Questionnaire | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kanwal Raghav, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org

DOCUMENTS (1):
  • Informed Consent Form (2021-05-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT05024968/ICF_000.pdf